CLINICAL TRIAL: NCT03213821
Title: Safety and Efficacy of High Protein Diet Versus Glomerular Filtration Rate (GFR) Based Protein Diet in Non-obese Advanced Heart Failure (HF) Patients With Renal Insufficiency: Randomized Controlled Trial
Brief Title: Safety and Efficacy of High Protein Diet Versus GFR Based Protein Diet in Heart Failure Patients With Renal Insufficiency
Acronym: GFR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 96001
Record Dates: First submitted 2017-05-08; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Study design A randomized, parallel-arm, controlled pilot study is designed. Sample size is determined 50 participants per treatment arm using the stepped rules of thumb, with standardized effect sizes of 0.1 or less and power 80% for main trial (n=100). After baseline assessments, balanced permuted block method will be used for randomization. Concealment of the randomization sequence will be performed by the RCT center of Rajaie Cardiovascular, Medical and Research Center. Intervention will be according to the randomization sequence.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high protein intake (Experimental): Study participants will receive high protein diet as recommended to preserve muscle mass (1.2-1.5 g/kg Ideal Body Weight)
  Interventions: Other: protein intake
- GFR based protein intake (Active Comparator): Study participants will receive GFR based protein diet to preserve renal function.
  Interventions: Other: protein intake

INTERVENTIONS:
Other: protein intake — For each participant, weighed food records of 3 consecutive days will be analyzed for estimation of calorie and macronutrient intake and dietary preferences. To make sure good compliance, diets will be developed regarding patient's dietary habits and preferences individually. High calorie (30-35 kcal/kg Ideal body weight) diets including 6-8 small meals will be formulated. Intervention group will receive high protein diet as recommended to preserve muscle mass (1.2-1.5 g/kg IBW). Comparison group will receive protein based on GFR to preserve renal function. For older adults (>65 years) protein content of diet will be as recommended by the international study group to review dietary protein needs with aging (PROT-AGE). In subjects with lower intake of protein, carbohydrate will be substituted. Both group will receive low fat diet.

SUMMARY:
Effect of high calorie high protein diet versus high calorie,glomerular filtration rate (GFR) based protein intake in non-obese advanced HF patients will be assessed. In this regard, protein intake impact will be measured on muscle mass, physical performance and renal function as main outcome. Rehospitalization, quality of life, depression an inflammatory status are second endpoints.

DETAILED DESCRIPTION:
Patient examinations:

Baseline data will be gathered on demographic and clinical characteristics, medical history, treatments and medications. Before initiating intervention, individuals will be assessed for anemia and 25 (OH) D2 and electrolytes status. Any insufficiency or imbalance will be corrected by drug therapy or supplementation. At baseline and at all visits, half or one month intervals, routine laboratory tests for heart failure patients (including Complete blood count (CBC), electrolytes status, glucose, albumin, cholesterol, triglyceride, blood urea nitrogen (BUN), C-reactive Protein (CRP),creatinine, uric acid, ferritin, 25 (OH) D, B-type natriuretic peptide (BNP), thyroid function, Prealbumin, urine analysis), appetite status and anthropometric measurements (weight, Hip and waist circumference) will be performed. At baseline and by the end of month 6, body composition, muscle mass, hand grip strength, Short Physical Performance Battery (SPPB), plasma lactate and interleukin 6 (IL-6), GFR, depression status and quality of life will be assessed. Follow up duration will be one year for measuring readmission and mortality rate. If a study participant did not attend a visit, a staff of randomized clinical trial (RCT) center will attempt to reach her/him, her/his designated friend or family member by phone call.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HF patients class III in New York Heart Association (NYHA) based on European Society of Cardiology (ESC) definition
* Hand grip strength less than normal for age,
* Age >18 years,
* Glomerular filtration rate (GFR) 30-90,
* BMI <30, muscle mass >2 standard deviations (SDs) below mean in individuals aged 18-39 y in the NHANES III cohort.

Exclusion Criteria:

* Respiratory failure,
* Ventilator dependence,
* Dialysis treatment, and sepsis,
* Open abdominal surgery within 6 weeks prior to enrolment,
* Diseases or conditions that might change the calorie and macronutrients requirement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline muscle mass at 6 months | At baseline and after 6 months
  muscle mass will be assessed by Dual-Energy X-Ray Absorptiometry (DEXA)

SECONDARY OUTCOMES:
Change from baseline depression status at 6 months | At Baseline and after 6 months
  Cardiac Depression Scale (CDS) questionnaire
Change from baseline appetite status at 6 months | At baseline, in each visit up to 6 months
  Simplified Nutritional Appetite Questionnaire (SNAQ)
Change from baseline quality of life status at 6 months | AT baseline and after 6 months
  Kansas City Cardiomyopathy Questionnaire
Mortality rate | Up to 1 year
  Mortality occurrence
Rehospitalization | Number of hospital admission will be recorded from date of intervention initiation until 1 year
  Frequency of hospital admission in 1 year
Change from baseline kidney function at 6 months | At baseline and after 6 months
  Glomerular filtration rate (GFR) (WIZARD® Automatic Gamma Counter) will be performed
Change from baseline handgrip strength at 6 months | At baseline and after 6 months
  Handgrip strength will be measured using hand grip dynamometer
Change from baseline physical performance at 6 months | At baseline and after 6 months
  SPPB score will be measured for physical performance assessment which includes: gait speed (timed 4-metre walk), sit-to-stand time (timed test of five chair rises), and standing balance (side-by-side stand, tandem and semi-tandem positions)

IPD SHARING:
Plan to Share IPD: No
Data will be kept confidential.